CLINICAL TRIAL: NCT04632147
Title: The Effect of Pranayamic Techniques on Obstructive Sleep Apnea Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Zeynep KAÇAR, physiotherapist, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 59491012-604.01.02
Record Dates: First submitted 2020-10-22; First posted 2020-11-17 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Obstructive Sleep Apnea Syndrome
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: Participants will be randomly divided into two groups as pranayama group and control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pranayama Group (Experimental): Participants in this group will apply a 45-minute training program at home, consisting of 5 minutes of Ujjayi pranayama, 5 minutes of Nadi-Shodhana pranayama and 5 minutes of Sukha pranayama, 7 days a week for 8 weeks, 3 times a day. In addition, they will perform a 15-minute session 3 day a week for 8 weeks, under the online supervision of a physiotherapist. The training program will last 8 weeks.
  Interventions: Other: Ujjayi pranayama, Nadi-Shodhana pranayama, Sukha pranayama
- Control Group (No Intervention): No intervention will be made to this group.

INTERVENTIONS:
Other: Ujjayi pranayama, Nadi-Shodhana pranayama, Sukha pranayama — Ujjayi pranayama:It is a pranayamic application that is performed by slightly twisting the throat and breathing through the nose. Nadi shodhana pranayama is breathing alternately through the right and left nostrils.Sukha pranayama is inhaled through the nose for 5 seconds, then given through the nose for 5 seconds. Thus, 6 times of inspiration and expiration is done per minute.
  Arms: Pranayama Group

SUMMARY:
Study was planned to investigate the effect of pranayama on dyspnea, daytime sleepiness, cognitive function, quality of life, activities of daily living, functional exercise capacity, physical activity level, sleep quality, fatigue, musculoskeletal pain, depression and anxiety in OSAS.

DETAILED DESCRIPTION:
Thirty-four OSAS patients meeting the inclusion criteria will be randomized into 2 groups as pranayama and control groups. The pranayama group will practice pranayama on their own for 8 weeks, 7 days a week, 3 times a day for 15 minutes. In addition, he will perform a single 15-minute session 3 days a week online under the supervision of a physiotherapist. The control group will not receive any intervention. Dyspnea sensation before and after the training Modified Medical Research Council dyspnea scale, daytime sleepiness Epworth Sleepiness Scale, cognitive function Montreal Cognitive Assessment Scale, quality of life Short Form-36, Turkish Adaptation of Nottingham Health Profile Questionnaire and Functional Outcomes of Sleep Questionnaire, activities of daily living London Chest Activities of Daily Living Scale, functional exercise capacity 30 seconds sit and stand test, physical activity level International Physical Activity Questionnaire-Short Form, sleep quality Pittsburgh Sleep Quality Index, fatigue status Fatigue Severity Scale, depression and anxiety Hospital Anxiety and Depression Scale, musculoskeletal system pain will be assessed with the Nordic Musculoskeletal Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with mild to moderate obstructive sleep apnea syndrome.

Exclusion Criteria:

* Using a mandibular advancement device
* Regularly using hypnotic drugs
* Have a metabolic disease (eg diabetes, hypothyroidism, obesity)
* Have Hypertension
* Have Malignancy
* Have Epilepsy
* Have Heart failure
* Have COPD
* Have asthma
* Neurological, psychological, cooperative problems
* Having a history of maxillofacial surgery

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2021-04-20 (Actual); Primary Completion 2021-09-20 (Estimated); Study Completion 2021-09-25 (Estimated)

PRIMARY OUTCOMES:
Vital Capacity | 8 weeks
  Vital capacity will be measured in liters, which is one of the respiratory functions.
Functional Exercise Capacity | 8 weeks
  It will be evaluated by the 6-minute walking test.
Dyspnoea | 8 weeks
  The resting dyspnea level will be evaluated according to the Modified Borg Scale.
fatigue | 8 weeks
  Fatigue level will be assessed using the Fatigue Severity Scale (FSS).
Anxiety and Depression Status | 8 weeks
  It will be evaluated with the Hospital Anxiety Depression Scale.
Physical Activity Level | 8 weeks
  It will be evaluated with the International Physical Activity Questionnaire-Short form (IPAQ-S).
Cognitive Function | 8 weeks
  Cognitive evaluation of the patients will be made with the Montreal Cognitive Assessment Scale (MOCA).
Daily Life Activities | 8 weeks
  Daily life activities will be evaluated with the London Chest Daily Living Activities Scale.
Daytime Sleepiness | 8 weeks
  Daytime sleepiness will be assessed with the Epworth Sleepiness Scale (ESS).
Sleep Quality | 8 weeks
  Sleep quality will be evaluated with the Pittsburg Sleep Quality Index (PSQI).
Life Quality | 8 weeks
  Quality of life will be evaluated with the SF-36 scale.
Inspiratory Muscle Strength | 8 weeks
  Inspiratory muscle strength will be evaluated by measuring the maximum inspiratory pressure (MIP) in cmH2O.
Forced Vital Capacity | 8 weeks
  Forced Vital Capacity will be measured in liters, which is one of the respiratory functions.
Expiratory Muscle Strength | 8 weeks
  Expiratory muscle strength will be evaluated by measuring the maximum expiratory pressure (MIP) in cmH2O.

CONTACTS AND LOCATIONS:
Overall Officials: Rengin Demir, Study Chair — Istanbul University Cerrahpasa Cardiology Institute; Ömer Önder Önder, Study Chair — Istanbul Esenyurt University Health Science Faculty; Ersan Atahan, Study Chair — Istanbul University Cerrahpasa Faculty of Medicine Department of Chest Diseases
Locations (1):
- Zeynep Kaçar, Istanbul, Türkiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Participants' age, gender, general health status, respiratory functions, functional exercise capacity, dyspnea level, fatigue severity, anxiety and depression status, physical activity level, cognitive function, daily living activities, daytime sleepiness, daily living activities, quality of life, respiratory muscle Data such as strength will be shared with other researchers. Other researchers will be able to obtain these data of the participants both before and after the intervention.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: starting 6 months after publication
Access Criteria: IPD will be shared with all researchers in the study.

REFERENCES:
- [Background] Armutlu K, Korkmaz NC, Keser I, Sumbuloglu V, Akbiyik DI, Guney Z, Karabudak R. The validity and reliability of the Fatigue Severity Scale in Turkish multiple sclerosis patients. Int J Rehabil Res. 2007 Mar;30(1):81-5. doi: 10.1097/MRR.0b013e3280146ec4. PMID 17293726
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Garrod R, Bestall JC, Paul EA, Wedzicha JA, Jones PW. Development and validation of a standardized measure of activity of daily living in patients with severe COPD: the London Chest Activity of Daily Living scale (LCADL). Respir Med. 2000 Jun;94(6):589-96. doi: 10.1053/rmed.2000.0786. PMID 10921765
- [Background] Polkey MI, Green M, Moxham J. Measurement of respiratory muscle strength. Thorax. 1995 Nov;50(11):1131-5. doi: 10.1136/thx.50.11.1131. No abstract available. PMID 8553266
- [Result] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893